CLINICAL TRIAL: NCT05661591
Title: Pharmacokinetic Effect of Fluconazole on SHR2554 in Healthy Subjects in Single-center, Open-label, Single-dose, Auto-controlled Pharmacokinetics
Brief Title: Effect of Fluconazole on Pharmacokinetics of SHR2554 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR2554-I-110
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms | interventions — Fluconazole

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, single-dose, self-control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group A (Experimental): SHR2554+ Fluconazole Capsules
  Interventions: Drug: SHR2554 Tablets; Drug: Fluconazole Capsules

INTERVENTIONS:
Drug: SHR2554 Tablets — SHR2554 Tablets+ Fluconazole Capsules
Drug: Fluconazole Capsules — SHR2554 Tablets+ Fluconazole Capsules

SUMMARY:
The study is being conduct to evaluate fluconazole effect of on SHR2554 in condition of single-canter, open-label, single-dose in healthy subjects. To explore the SHR2554 pharmacokinetics change under use of fluconazole and insure the safety with SHR2554 combined with fluconazole.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial, fully understand the trial process and possible adverse reactions in trail, and be able to complete the research in accordance with the requirements of the trail protocol;
2. Healthy male and female subjects aged 18 to 45 year the date of signing the informed consent form, with female subjects ratio is not less than 40%;
3. Male subjects weighed ≥ 50kg, female subjects weighed ≥ 45kg, and body mass index (BMI) was in the range of 19.0~26.0kg/m2 (including the cut-off value);
4. No family plan for the next 30 days and voluntary use of highly effective contraception during the trial.

Exclusion Criteria:

1. Allergies, including severe drug allergies or drug allergies; history of allergy to SHR2554 tablets, fluconazole capsules, or their excipients;
2. A clear history of primary diseases of important organs such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolic and musculoskeletal system, including but not limited to tumour patients or tumour history, which the investigator believes is not suitable to participate in this study;
3. During screening, comprehensive physical examination, vital signs examination (breathing, blood pressure, pulse and body temperature), chest orthostatic X-ray, and laboratory tests (blood biochemistry, blood routine, urine routine, immunization eight, coagulation function, female pregnancy) and other abnormal clinical significance (subject to the judgment of the clinician);
4. Screening of male QTcF ≥ 430 msec or female QTcF ≥ 450 msec by electrocardiogram examination, or abnormal clinical significance judged by the investigator in the ECG results;
5. Have a history of drug and/or alcohol abuse, positive alcohol and drug screening, or have a history of drug abuse within the past five years or have used drugs in the 3 months before the trail;
6. Addicts to tobacco and alcohol (drinking ≥ 14 units of alcohol per week) in the 3 months before screening: 1 unit = 360mL of beer, or 45mL of spirits, or 150mL of wine; Those who smoke ≥5 cigarettes) daily and cannot ban smoking and alcohol during the test;
7. Those who have undergone any surgery within 6 months before screening;
8. Hepatotoxic drugs (such as itraconazole, dapsone, erythromycin, fluconazole, ketoconazole, rifampicin, isoniazid, tetracycline, glibenclamide, propylthiouracil, methimazole, statin lipid-lowering drugs, fenofibrate, etc.) within 6 months before screening;
9. Use of any drugs that alter the activity of CYP3A enzyme (such as carbamazepine, phenytoin, modafinil, ritonavir, voriconazole, St. John's wort, bosentan tablets, efavirenz, etravirine, ciprofloxacin, etc.) within 28 days before taking the study drug;
10. Use of any prescription drug, over-the-counter drug, vitamin product, supplement or herbal medicine within 14 days before taking the trail drug;
11. ingested grapefruit or grapefruit-containing products, caffeinated, xanthine, or alcoholic foods or beverages within 48 hours prior to taking the study drug; strenuous exercise, or other factors that affect drug absorption, distribution, metabolism, excretion and other factors;
12. Those who participated in blood donation within 3 months before taking the study drug and donated blood ≥ 200mL, or received blood transfusion;
13. Those with a history of needle sickness and blood sickness, difficulty in blood collection or inability to tolerate venous puncture blood collection;
14. female subjects lactating; Male subjects who have a sperm donation plan from the signing of the informed consent form until 30 days after the last dose of the experimental drug;
15. Those who have participated in other drug trials within 3 months before screening;
16. participants who the investigator believes have other factors that are not suitable for participation in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of SHR2554: Cmax | day 1 to day 10
Pharmacokinetic parameters of SHR2554: AUC0-t | day 1 to day 10
Pharmacokinetic parameters of SHR2554: AUC0-∞ | day 1 to day 10

SECONDARY OUTCOMES:
Pharmacokinetic parameters of SHR2554: Tmax | day 1 to day 10
Pharmacokinetic parameters of SHR2554: t1/2 | day 1 to day 10
Pharmacokinetic parameters of SHR2554: CL/F | day 1 to day 10
Pharmacokinetic parameters of SHR2554: Vz/F | day 1 to day 10
The incidence and severity of adverse events/serious adverse events | from ICF signing date to approximate day 18

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided